CLINICAL TRIAL: NCT02218619
Title: Clinical Investigation of Efficacy of Tauroursodeoxycholic Acid (TUDCA) to Enhance Pancreatic Beta Cell Survival In Type 1 Diabetes by Reducing Endoplasmic Reticulum Stress
Brief Title: Tauroursodeoxycholic Acid (TUDCA) in New-Onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robin Goland, MD (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Robin Goland, MD, J. Merrill Eastman Professor of Clinical Diabetes, Co-Director, Berrie Center, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAN2402
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes (T1D); endoplasmic reticulum (ER) stress; induced pluripotential stem (iPS) cells; Tauroursodeoxycholic Acid (TUDCA)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Ichthyosis prematurity syndrome | interventions — ursodoxicoltaurine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taurourodeoxycholic Acid (TUDCA) (Experimental): TUDCA 1750 mg/day x 12 months
  Interventions: Drug: Tauroursodeoxycholic Acid (TUDCA)
- Sugar pill (placebo) (Placebo Comparator): Placebo at same dose, frequency, and duration as experimental treatment
  Interventions: Drug: Sugar Pill (placebo)

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid (TUDCA) — TUDCA at 1750 mg/day x 12 months
  Other Names: TUDCA; Taurolite
  Arms: Taurourodeoxycholic Acid (TUDCA)
Drug: Sugar Pill (placebo) — Placebo
  Other Names: Placebo
  Arms: Sugar pill (placebo)

SUMMARY:
Clinically, the ability to slow or prevent beta cell demise can prevent or improve the course of type 1 diabetes. The immune-mediated destruction of beta cells that is an apparent major pathological basis for the disease, has led to efforts to prevent or suppress this immune assault. Here the investigators propose to buttress the beta cell's capacity to withstand this assault by improving the function of the endoplasmic reticulum stress resolving mechanisms within these cells. The ability to do so could have a major impact on preventive and therapeutic strategies for type 1 diabetes (and possibly other types of diabetes). The type of endoplasmic reticulum stress relieving agent (TUDCA) proposed here could ultimately be applied on an anticipatory basis to individuals at high risk for type 1 diabetes.

DETAILED DESCRIPTION:
Reducing endoplasmic reticulum stress will promote beta cell survival in new-onset type 1 diabetes.

The primary aim is to test the clinical efficacy of an already approved agent, TUDCA, re-purposed to reduce endoplasmic reticulum stress and improve beta cell survival in patients with new onset type 1 diabetes. The primary endpoint of this proposed double-blinded randomized placebo-controlled pilot study is c-peptide measured after mixed meal stimulation test at randomization and then at 6 and 12 months of treatment with TUDCA compared to treatment with placebo and at 6 months following treatment.

TUDCA is an oral medication with a safety profile that is approved for use in Europe for gall stones and liver disease. The drug and similar compounds has been used in children, as young as newborns, and in adults. TUDCA's ability to lower endoplasmic reticulum stress has only recently been recognized and will be applied to new-onset type 1 diabetes in this proposal. If this pilot trial is successful, future studies could include broadening the recipients to antibody-positive pre-type 1 diabetes patients and/or combining TUDCA with other agents shown to have a beneficial effect on insulin secretion in new-onset type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to American Diabetes Association criteria
* Diagnosis of type 1 diabetes within 100 days of randomization
* One positive diabetes-related autoantibody
* Ages 18-45 years

Exclusion Criteria:

* Drugs known to affect glucose other than insulin
* Stimulated C-peptide levels < 0.2 pmol/ml measured during a mixed meal tolerance test conducted at least 21 days from diagnosis of diabetes and within one month (37 days) of randomization to either TUDCA or placebo.
* Women during pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Goland, MD, Principal Investigator — Columbia University; Rudolph Leibel, MD, Principal Investigator — Columbia University
Locations (1):
- Naomi Berrie Diabetes Center, Columbia University, 1150 St. Nicholas Ave., New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
primary data to be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2021
Access Criteria: email rsg2@columbia.edu

REFERENCES:
- [Derived] Rosa LRO, Vettorazzi JF, Zangerolamo L, Carneiro EM, Barbosa HCL. TUDCA receptors and their role on pancreatic beta cells. Prog Biophys Mol Biol. 2021 Dec;167:26-31. doi: 10.1016/j.pbiomolbio.2021.09.003. Epub 2021 Sep 20. PMID 34547326

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taurourodeoxycholic Acid (TUDCA) | Sugar Pill (Placebo)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Glutamic acid decarboxylase (GAD) Result [Count of Participants; unit: Participants]
  GAD Negative | 0 | 1 | 1
  GAD Positive | 10 | 9 | 19
Islet cell antigen 2 (IA2) Result [Count of Participants; unit: Participants]
  IA2 Negative | 7 | 3 | 10
  IA2 Positive | 3 | 7 | 10
Insulin Autoantibodies (IAA) Result [Count of Participants; unit: Participants]
  IAA Negative | 5 | 5 | 10
  IAA Positive | 5 | 5 | 10
Pancreatic islet-cell antibodies (ICA) Result [Count of Participants; unit: Participants]
  ICA Negative | 4 | 1 | 5
  ICA Positive | 6 | 9 | 15
Zinc Transporter 8 Autoantibody (ZnT8A) Result [Count of Participants; unit: Participants]
  ZnT8A Negative | 4 | 4 | 8
  ZnT8A Positive | 6 | 6 | 12
Positive Autoantibodies [Mean (Standard Deviation); unit: Positive Autoantibodies] | 3 (1.49) | 3.6 (1.17) | 3.3 (1.34)
Days from Diagnosis to Randomization [Mean (Standard Deviation); unit: Days] | 87.50 (47.44) | 67.70 (21.41) | 77.60 (37.24)
Weight [Mean (Standard Deviation); unit: Kilograms] | 72.50 (10.18) | 69.05 (9.17) | 70.78 (9.59)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.91 (2.85) | 23.26 (2.86) | 24.09 (2.91)
Area Under Curve (AUC) for C-Peptide [Mean (Standard Deviation); unit: nmol/L*120 min] | 0.53 (0.20) | 0.54 (0.27) | 0.53 (0.23)
Hemoglobin A1C (HbA1C) [Mean (Standard Deviation); unit: Percent] | 7.10 (0.95) | 8.65 (2.19) | 7.88 (1.83)
Total Daily Insulin Dose (Average 3 days before baseline visit) [Mean (Standard Deviation); unit: units/kg] | 0.22 (0.12) | 0.40 (0.16) | 0.31 (0.17)

OUTCOME MEASURES:

1. Primary Outcome: Change in C-peptide Measurement as Reflection of Insulin Secretion at 6 Months
Description: The primary endpoint will be the change from baseline in area under the stimulated C-peptide curve over the first 2 hours of a 4- hour mixed meal tolerance test conducted at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: nmol/L*120 min
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
nmol/L*120 min | -0.07 (0.11) | -0.07 (0.10)

2. Primary Outcome: Change in C-peptide Measurement as Reflection of Insulin Secretion at 12 Months
Description: The primary endpoint will be the change from baseline in area under the stimulated C-peptide curve over the first 2 hours of a 4- hour mixed meal tolerance test conducted at 12 months.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: nmol/L*120 min
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
nmol/L*120 min | -0.10 (0.18) | -0.12 (0.17)

3. Primary Outcome: Change in C-peptide Measurement as Reflection of Insulin Secretion at 18 Months
Description: The primary endpoint will be the change from baseline in area under the stimulated C-peptide curve over the first 2 hours of a 4- hour mixed meal tolerance test conducted at 18 months
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: nmol/L*120 min
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
nmol/L*120 min | -0.11 (0.21) | -0.14 (0.16)

4. Secondary Outcome: Number of Participants With Liver Function Test Abnormalities
Description: Measure liver function tests at 6 and 12 months and at 6 months after drug or placebo is stopped to ensure that no abnormalities (liver function blood tests outside of normal reference range) of liver function occur with the drug.
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
Participants
  Month 6 | 0 | 0
  Month 12 | 0 | 0
  Month 18 | 0 | 0

5. Secondary Outcome: Change in Insulin Use at 6 Months
Description: Change in insulin use from baseline at 6 months
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
units/kg | -0.10 (0.18) | 0.09 (0.23)

6. Secondary Outcome: Change in Insulin Use at 12 Months
Description: Change in insulin use from baseline at 12 months
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
units/kg | -0.10 (0.14) | 0.09 (0.16)

7. Secondary Outcome: Change in Insulin Use at 18 Months
Description: Change in insulin use from baseline at 18 months
Time Frame: Baseline and 18 months
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
units/kg | -0.17 (0.18) | 0.02 (0.21)

8. Secondary Outcome: Change in HbA1c at 6 Months
Description: Change in HbA1c from baseline at 6 months
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
Percent | -0.98 (1.57) | -2.27 (2.13)

9. Secondary Outcome: Change in HbA1c at 12 Months
Description: Change in HbA1c from baseline at 12 months
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
Percent | -0.02 (3.31) | -2.25 (2.13)

10. Secondary Outcome: Change in HbA1c at 18 Months
Description: Change in HbA1c from baseline at 18 months
Time Frame: Baseline and 18 Months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 10 | 10
Percent | -0.48 (2.22) | -1.89 (2.14)

11. Other Pre Specified Outcome: Endoplasmic Reticulum Stress
Description: It is believed that the autoimmune assault of new onset type 1 diabetes leads to stress to the part of the beta cell that folds proteins; referred to as endoplasmic reticulum stress. When endoplasmic reticulum stress increases, changes in protein levels in beta cells occur. The investigators will measure markers of endoplasmic reticulum stress in beta cells taken from skin biopsies from subjects before treatment with TUDCA or placebo.
Time Frame: 1 week
Population: Biopsy samples were collected, but not sent for pathological analysis due to trial futility. There are no results available to report.
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Sugar Pill (Placebo) | Taurourodeoxycholic Acid (TUDCA)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02218619/Prot_SAP_000.pdf